CLINICAL TRIAL: NCT00719745
Title: A Phase III, Randomized, Open-Label, Comparative, Multi-Center Study to Assess the Safety and Efficacy of Prograf® (Tacrolimus) and MR4 (Modified Release Tacrolimus) in de Novo Liver Transplant Recipients
Brief Title: A Study to Assess the Safety and Efficacy of Prograf and MR4 in Liver Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Director, Astellas Pharma Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-05-02-KOR
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Liver Transplantation
Keywords: Organ transplantation; Tacrolimus; Prograf; MR4
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Prograf
- 2 (Experimental)
  Interventions: Drug: MR4

INTERVENTIONS:
Drug: Prograf — oral
  Other Names: Tacrolimus; FK506
  Arms: 1
Drug: MR4 — oral
  Other Names: Modified Release Tacrolimus; FK506MR; FK506E
  Arms: 2

SUMMARY:
To evaluate and to compare efficacy and safety of MR4 versus Prograf in patients undergoing primary liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of child bearing potential must have a negative in pregnancy test prior to enrollment and must agree to practice effective birth control during the study
* Patients who need liver transplantation due to the end-stage liver failure

Exclusion Criteria:

* Patients receiving multi-organ transplant or having previously received an organ transplant ( including re-transplantation)
* Patients receiving auxiliary graft or in whom a bio-artificial
* Patients allergic to macrolide antibiotics or tacrolimus
* Patients requiring immunosuppressive treatment or systemic chemotherapy prior to transplantation. Patients requiring low level immunosuppressive treatment ( MMF, steroids, azathioprine ) before transplantation to control their original liver disease can be included in the study, provided that this treatment is discontinued at the time of transplantation. Local chemotherapy is allowed
* Patients with malignancies of a history of malignancy within the last 5 years, with the exception of those with basalioma or squamous cell carcinoma of the skin that has been treated successfully Patients can be included under Milan Criteria Patients with malignancy which was identified after completion of surgery e.g. by histopathology will be allowed to remain in the study
* Patients with systemic infection requiring treatment, except viral hepatitis
* Patients with severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patients with serum creatinine > 1.5mg/Dl
* Patients with any form of substance abuse, psychiatric disorder of condition which, in the opinion of the investigator, may complicate communication with the investigator
* Patients participating or participated in another clinical trial or those taking or having taken an investigational / non-registered drug in the past 28 days
* Patients who are pregnant or breast-feeding mother
* Patients or donors known to be HIV positive
* Patients unlikely to comply with the visits scheduled in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Event rate of patients with biopsy-proven acute rejections | 24 weeks

SECONDARY OUTCOMES:
Incidence of and time to acute rejections and corticosteroid resistant acute rejections | 12 and 24 weeks
Severity of biopsy-proven acute rejections. | 24 weeks
Patient and graft survival | 12 and 24 weeks
Incidence of adverse events | Throughout trial

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Korea, Inc.
Locations (1):
- Seoul, South Korea